CLINICAL TRIAL: NCT05582915
Title: Screening for Prognostic Biomarkers of Severe Bell's Palsy in Adults Using Proteomic Analysis by Quantitative Mass Spectroscopy
Brief Title: Screening for Prognostic Biomarkers of Severe Bell's Palsy in Adults
Acronym: BIOFIPS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0036
Record Dates: First submitted 2022-10-05; First posted 2022-10-17 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Bell Palsy
Keywords: Bell's palsy; Proteomics; Biomarkers; Mass spectroscopy; Prognosis
MeSH Terms: conditions — Bell Palsy | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma collection for proteomic analysis (after veinous blood centrifugation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with severe Bell's palsy: Adult patients recently diagnosed with severe Bell's palsy and referred to the ENT Department by A&E or by general practitionner.
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — 4 ml of blood will be collected into EDTA tube for proteomic analysis at visit 0 and visit 1

SUMMARY:
Bell's palsy (idiopathic peripheral facial palsy) is the most common cause of facial palsy, which is related to the inflammation of the facial nerve, possibly induced by herpesvirus reactivation. Its first-line treatment comprises corticosteroids, antiviral therapy and physiotherapy. In most severe cases (grade IV to VI on House-Brackmann scale), facial motricity may remain altered or develop synkinesis or post-paralytic spasm, thus tremendously affecting quality of life. To avoid potential complications, surgical facial nerve decompression could be proposed. To date, however, there are no means to predict if Bell's palsy will evolve with any complications or if the patient will recover entirely. Thus, the invasive facial nerve decompression is equally proposed to subjects who will develop the consequences as well as to subjects able to restore without surgical treatment. This study proposes to search for prognostic blood biomarkers related to the Bell's palsy recovery pattern. Adult patients with severe Bell's palsy will be proposed to have a blood sampling for proteomic analysis in the early stage of the disease. Then 125 biomarkers on a Peptiquant™ kit will be analysed by mass spectrometry, and prognostic biomarkers will be selected regarding to the clinical recovery of Bell's palsy

DETAILED DESCRIPTION:
Bell's palsy (idiopathic peripheral facial palsy) is the most common cause of facial palsy, which is related to the inflammation of the facial nerve, possibly induced by herpesvirus reactivation. Its first-line treatment comprises corticosteroids, antiviral therapy and physiotherapy. In most severe cases (grade IV to VI on House-Brackmann scale), facial motricity may remain altered or develop synkinesis or post-paralytic spasm, thus tremendously affecting quality of life. The recovery of Bell's palsy is currently evaluated either by Sunnybrook Facial Grading System, House-Brackmann scale or Chevalier's method. It is nonetheless unpredictable, especially at the early stage of the disease.

If the first-line treatment fails to provide a fast recovery, facial nerve decompression surgery may be proposed. Being rather complex and risky, this technique shows a lower efficiency if delayed from the onset. Surgical indication is based upon clinical and radiological criteria as well as electrophysiological measurements (electromyography - EMG and electromyoneurography - EMNG). EMG and ENMG methods have a somewhat limited predictive value, since 20 to 40% patients with severe Bell's palsy can recover without surgical treatment. Moreover, these measurements are not widely accessible and, in severe cases, they should be performed between 9 and 20 days from the onset. The surgery, in order to increase its success rate, should be performed in maximum 30 days, ideally in 14 days from the onset.

Therefore, diagnostic and treatment of severe Bell's palsy face a double challenge: a narrow time window to provide a diagnostic and therapeutic strategy, and the need of a reliable prognostic methods to exclude the possibility of spontaneous recovery and thus to justify the surgical approach.

Mass Spectrometry assay allows simultaneous detection of numerous proteins, to screen for inflammatory and neurodegenerative biomarkers at acute stage of Bell's palsy. Some of these proteins might appear of a prognostic value and will help to develop more reliable and personalised treatment approach of severe Bell's palsy.

The primary objective of the study is to identify prognostic blood biomarkers related to the facial motricity recovery at 3 months from onset of severe Bell's palsy in adults.

The secondary objectives are identification of the biomarkers related to the recovery speed in the first three months, and to the initial severity of Bell's palsy; evaluation of diagnostic performance of selected biomarkers; creation of a blood collection for further research on selected biomarkers.

130 patients referred by accident and emergency department will be enrolled during their appointments at the ENT Department of the University Hospital of Montpellier. BIOFIPS study implies 4 visits, with the overall duration of 3 months per patient. After patient information and consent, routine clinical examination, audiometric testing, tympanometry, acoustic reflex testing and Bell's palsy scoring will be performed. Patients will receive a medical prescription for a blood test an MRI to exclude other causes of facial palsy. At time of inclusion and 1 month after, they will be proposed to have a blood sampling for proteomic analysis. Then 125 biomarkers on a Peptiquant™ kit will be analysed by mass spectrometry, and prognostic biomarkers will be selected regarding to the clinical recovery of Bell's palsy.

ELIGIBILITY:
Inclusion Criteria:

* Severe Bell's palsy (House-Brackmann more or equal to IV)
* Disease developed between 5 and 15 days before V0 (after initial corticotherapy)
* 18 years and older

Exclusion Criteria:

* Facial palsy (central or peripheral) of a following cause suspected at V0:

Diabetes, syphilis, HIV-1 or HIV-2 infection, Lyme disease, herpes zoster infection of the geniculate ganglion; Inflammatory or immune pathology, acute or chronic; Intracranial, parotid or facial nerve tumor; Craniofacial injury; Other peripheral neuropathy

* Anti-inflammatoty, immunomodulating, immunosuppressive treatment
* Contraindications for an MRI scan
* Contraindications for a standard medical treatment: prednisone 1 mg per kg a day during 5 days and valaciclovir 3 g a day during 7 days
* Contraindications for or an impossibility of facial physiotheraphy (2 times per week along with everyday self-theraphy)
* Pregnancy or breastfeeding
* Participation to another interventional study
* Patient unaffiliated to French Social Security regime
* Patients' refusal to consent to participation in the study
* Person prived of liberty by judicial or administrative decision
* Person protected by law (under guardianship or curatorship)
* Person not able to understand the nature, the aim and the methodology of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults recently diagnosed with severe Bell's palsy and referred to the ENT department by A&E or general practitionner.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Area under the ROC curve of biomarkers (from initial sampling) for prognosis of facial motricity recovery at 3 months | Visit 0, Visit 1, Visit 2 and Visit 3 (3 months)
  "no recovery" group: gain (Visit 3-Visit 0) <40% on Chevalier score vs. "recovery" group: gain (Visit 3-Visit 0) ≥40% on Chevalier score.
  Chevalier score is a clinical scale that evaluates the percentage of facial motricity regarding 15 facial muscles.

SECONDARY OUTCOMES:
Biomarkers related to the speed of recovery in the first 3 months | Visit 0, Visit 1, Visit 2 and Visit 3
  Biomarkers (value or kinetic between Visit 0 and Visit 1 samples) related to the speed of recovery in the first 3 months: no recovery vs. recovery of PFPI
Biomarkers related to the initial severity of Bell's palsy | Visit 0
  Biomarkers at Visit 0 related to the initial severity of Bell's palsy (House and Brackmann score): HB IV vs. IPF HB V vs. IPF HB VI
Diagnostic value of selected biomarkers | Visit 0, Visit 1, Visit 2 and Visit 3
  specificity, positive and negative predictive value

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France